CLINICAL TRIAL: NCT00929019
Title: mRNA Transfected Dendritic Cell Vaccination in High Risk Uveal Melanoma Patients
Brief Title: Messenger Ribonucleic Acid (mRNA) Transfected Dendritic Cell Vaccination in High Risk Uveal Melanoma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rotterdam Eye Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL22553.000.08; KUN2008-035
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2015-09

CONDITIONS: Uveal Melanoma
Keywords: uveal melanoma; chromosome 3; high risk; immunotherapy; adjuvant; high risk genetic profile; loss of chromosome 3
MeSH Terms: conditions — Uveal Melanoma | interventions — RNA, Messenger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dendritic cell vaccination (Experimental): HLA-A2.1 positive patient will receive 3 biweekly intradermal/intravenous vaccination with autologous mRNA transfected mature dendritic cells, followed by a DTH skin test for monitoring purposes. One such cycle is repeated every 6 months if no signs of progression, up to a total of 3 cycles.
  Interventions: Biological: autologous dendritic cells electroporated with mRNA
- control arm (No Intervention): For comparison, HLA-A2.1 negative patients will be monitored for clinical response (secondary endpoint).

INTERVENTIONS:
Biological: autologous dendritic cells electroporated with mRNA — Autologous mature monocyte-derived dendritic cells electroporated with mRNA encoding gp100 and tyrosinase are vaccinated intradermal/intravenously 3 times with biweekly intervals every 6 months, if no signs of progression, for a total of 9 vaccinations.
  Arms: dendritic cell vaccination

SUMMARY:
1. Rationale

   Immunotherapy applying ex vivo generated and tumor antigen-loaded dendritic cells (DC) has now successfully been introduced in the clinic. A limited, but consistent, number of objective immunological and clinical responses have been observed. Most of the successful results have been observed in patients with minimal residual disease, rather than patients with advanced metastatic disease. Moreover, the investigators' preliminary results show that presence of tumor epitope specific T cells in biopsies taken from delayed type hypersensitivity (DTH) reaction sites highly correlates with prolonged progression free survival (PFS).

   Within uveal melanoma patients, a group with high risk of metastatic disease can be identified on basis of tumor specific genetic changes in loss of chromosome 3.

   At present no standard adjuvant or systemic treatment is available. Applying DC-based immunotherapy in this group of high risk patients might reduce the risk of recurrence without interference in the current treatment guidelines.
2. Objectives

   In this joint clinical study of Radboud University Nijmegen Medical Centre (RUNMC) and Rotterdam Eye Hospital, the investigators aim to determine the in vivo immunological response induced in high risk uveal melanoma patients vaccinated with mRNA-transfected DC.
3. Study design

   This study is an open label non-randomized phase II intervention study.
4. Study population

   The investigators' study population consists of HLA-A2 positive patients with a high risk uveal melanoma with proven expression of melanoma associated antigens tyrosinase and/or gp100.
5. Main study endpoints

This is an exploratory study aiming to demonstrate proof of principle. The first study endpoints are in vivo immunological response induced in high risk uveal melanoma patients vaccinated with mRNA-transfected DC, administered i.v./i.d. and toxicity. Secondary study endpoints are progression free survival, overall survival, and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* histological documented uveal melanoma
* HLA-A2.1 phenotype (intervention arm)
* non-HLA-A2.1 phenotype (control arm)
* melanoma expressing gp100 and/or tyrosinase
* high risk genetic profile (loss of chromosome 3) determined by FISH
* interval since local treatment of uveal melanoma < 12 months
* no signs of liver metastasis determined by diagnostic CT-abdomen
* normal serum LDH
* no signs of cerebral metastases
* bilirubin < 25 micromol/l
* WHO performance scale 0-1
* age 18-75 years
* written informed consent
* expected adequacy of followup
* no pregnant or lactating women

Exclusion Criteria:

* history of second malignancy, except adequately treated basal cell carcinoma
* serious active infections
* autoimmune disease or organ allografts
* concomitant use of immunosuppressive drugs
* known allergy to shell-fish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
immunological response | 2 years

SECONDARY OUTCOMES:
clinical response (progression free survival) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis JA Punt, prof.MD, Principal Investigator — Radboud University Nijmegen Medical Centre, Dept of Medical Oncology
Locations (2):
- Netherlands (2):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - The Rotterdam Eye Hospital, Rotterdam, South Holland

REFERENCES:
- See also: Radboud University Nijmegen Medical Centre — http://www.umcn.nl/Pages/default.aspx
- See also: Rotterdam Eye Hospital — http://www.oogziekenhuis.nl